CLINICAL TRIAL: NCT02308605
Title: A Field Deployable Blood Test for Stroke, Capable of Detecting Brain Ischaemia From the Earliest Stages of Pathology
Brief Title: SMARTCap Stroke Study: A Field Deployable Blood Test for Stroke
Acronym: SMARTCAP
Status: Completed | Type: Observational
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Responsible Party: Principal Investigator, Professor Christopher Imray, Professor Christopher Imray, Consultant Vascular Surgeon, University Hospitals Coventry and Warwickshire NHS Trust
Other Study IDs: CI126414 23 May 2014 V1; NIHR (Other Grant/Funding Number: ll-LA-0313-20002)
Record Dates: First submitted 2014-10-03; First posted 2014-12-04 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Stroke
Keywords: SMARTCap
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Suspected stroke patients and subset: Blood samples taken on admission and at 24 hours, MRI scan between 24 and 48 hours
  Subset: Blood samples repeated once per hour for six hours
  Interventions: Device: SMARTCap
- Control participants (relatives): To donate blood on two occasions, 24 hours apart, to draw comparison with stroke patients
  Interventions: Device: SMARTCap
- Feeding control participants: To donate a baseline blood sample, eat a simple purine rich meal (meat sandwich), then donate 4 more blood samples at 10, 30, 60 and 120 minutes following the meal
  Interventions: Device: SMARTCap

INTERVENTIONS:
Device: SMARTCap — The Sarissa Biomedical SMARTCap biosensor array. This is an array of biosensors and electrodes in a simple moulded device that will fit into a vacutainer blood tube and will enable the rapid measurement of purines in freshly drawn blood. Therefore, this is not an intervention as such as the device is an In-Vitro Diagnostic Medical Device.

SUMMARY:
The hypothesis is that a stroke causes release of purines from brain into blood and that this is a very early biomarker of brain ischaemia. The investigators propose a simple blood test of substances (the purines) that result from cellular metabolism and are produced in excess when brain cells are starved of oxygen and glucose (as occurs during a stroke).

DETAILED DESCRIPTION:
In this study, the investigators propose to use newly developed biosensor technology (SMARTCap) to directly address whether purines are indicators of real strokes, and can distinguish strokes from other conditions with similar symptoms, more rapidly.

ELIGIBILITY:
Inclusion Criteria:

1. Stroke patients: Admitted to the Hyperacute Stroke Unit having a suspected stroke within 1 hour of admission. Important to note that not all these patients will have suffered a stroke
2. Control participants: Relatives of patients admitted to the stroke treatment pathway, who are healthy and have no signs of cardiovascular illness
3. Healthy volunteers

Exclusion Criteria:

1. Stroke patients: Delay in admission exceeds the time window of 4 hours between stroke symptoms and admission
2. Control participants: Obvious signs or history of cerebrovascular disease
3. Unhealthy volunteers

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 320
Sampling Method: Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2014-09; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
To measure the levels of purine in the blood in Stroke patients compared to non-stroke patients (Healthy controls) | 30 minutes down to 5 minutes

SECONDARY OUTCOMES:
To identify ischaemic versus haemorrhagic strokes by combining purine measurements and CT scans | 24 hours to 7 days

OTHER OUTCOMES:
To measure the change in purines and their variability in control patients from baseline to day 7 | 24 hours - 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Christopher HE Imray, MB BS FRCP PhD, Principal Investigator — University Hospitals Coventry & Warwickshire NHS Trust
Locations (2):
- United Kingdom (2):
  - University Hospitals Coventry & Warwickshire NHS Trust, Coventry
  - University of Keele, Stoke-on-Trent

REFERENCES:
- [Derived] Dale N, Tian F, Sagoo R, Phillips N, Imray C, Roffe C. Point-of-care measurements reveal release of purines into venous blood of stroke patients. Purinergic Signal. 2019 Jun;15(2):237-246. doi: 10.1007/s11302-019-09647-4. Epub 2019 Mar 12. PMID 30859371